CLINICAL TRIAL: NCT03702491
Title: A Single-center Open, Randomized, Controlled Study to Compare the Apapitatin Combined With SOX and SOX for Palliative Adjuvant Chemotherapy in Patients With Advanced Gallbladder Carcinoma
Brief Title: Apapitatin Combined With SOX for Palliative Adjuvant Chemotherapy in Patients With Advanced Gallbladder Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Xiaoqing Jiang, Professor Chief Physician, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJiang
Record Dates: First submitted 2018-10-07; First posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-08

CONDITIONS: Gallbladder Carcinoma
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — apatinib; Tegafur; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib with SOX(Tegafur,Oxaliplatin) (Experimental): Patients 3-4 weeks after surgery, the SOX regimen was given palliative adjuvant chemotherapy for 6-8 cycles, then followed by the second cycle combined with the treatment of apatinib mesylate and the monotherapy maintenance of apatinib mesylate
  Interventions: Drug: Apatinib
- SOX( Tegafur,Oxaliplatin) (Active Comparator): 3-4 weeks after operation, 6-8 cycles of adjuvant chemotherapy with simple SOX protocol were given.
  Interventions: Drug: Tegafur

INTERVENTIONS:
Drug: Apatinib — Three to four weeks after surgery, the SOX regimen was given palliative adjuvant chemotherapy for 6-8 cycles, then followed by the second cycle combined with the treatment of apatinib mesylate and the monotherapy maintenance of apatinib mesylate
  Other Names: Tegafur; Oxaliplatin
  Arms: Apatinib with SOX(Tegafur,Oxaliplatin)
Drug: Tegafur — 3-4 weeks after operation, 6-8 cycles of adjuvant chemotherapy with simple SOX protocol were given.
  Other Names: Oxaliplatin
  Arms: SOX( Tegafur,Oxaliplatin)

SUMMARY:
A Single-center Open, Randomized, Controlled Study to Compare the Apapitatin Mesylate Combined With SOX Regimen and SOX Regimen for Palliative Adjuvant Chemotherapy in Patients With Advanced Gallbladder Carcinoma

DETAILED DESCRIPTION:
The aim of the study is to observe and evaluate the progression-free survival time (PFS), overall survival time (OS) and safety of patients with advanced Gallbladder Carcinoma treated with apatinib mesylate combined with SOX

ELIGIBILITY:
Inclusion Criteria:

1. ages 18 to 75
2. UICC/AJCC gallbladder TNM staging (The eighth edition), Ⅲ B - ⅣB (excluding M1) postoperative pathological diagnosis of gallbladder carcinoma;Patients confirmed to have undergone R1/R2 cholecystectomy or palliative surgery;
3. The primary treatment is surgical resection or potentially resectable cholecystic carcinoma without other treatment
4. ECOG performance status ≤1
5. The liver and kidney function meets the following conditions： BIL<3 normal value upper limit (ULN)；ALT and AST< 2.5 xULN;Serum Cr≤ 1xULN,Clearance rate of endogenous creatinine>50ml/min（Cockcroft-Gault）;
6. Other test rooms meet the following requirements:

   Hemoglobin ≥ 90 g/L (no blood transfusion within 14 days)；Neutrophilic granulocyte count > 1.5x109 /L;The platelet count ≥ 80 x 10 ^ 9/L;
7. Estimated life expectancy > 3 months.
8. Before the enrollment, the heart function is good. There is no episode of myocardial infarction within half a year. For example, if you have hypertension or coronary heart disease, you should ensure that it is within the controllable range.
9. Patient able and willing to provide written informed consent and to comply with the study protocol and Good compliance, with follow-up.

Exclusion Criteria:

1. Non gallbladder carcinoma
2. Significant clinical bleeding symptoms or a clear tendency to bleed occurred within the first month of randomization, such as cough/hemoptysis of 2.5ml or more, gastrointestinal bleeding, esophagogastric varices at risk of bleeding, hemorrhagic gastric ulcer, etc.
3. Other topical treatments during the study (including intraperitoneal chemotherapy, radiotherapy, etc.)
4. Pregnant or lactating women；
5. Those who suffer from high blood pressure and cannot be treated to the normal range by antihypertensive drugs；
6. HIV infection or the presence of AIDS-related diseases, or severe acute and chronic diseases;
7. Have grade II or higher myocardial ischemia or myocardial infarction、Poorly controlled arrhythmia；
8. Severe active infections；
9. There are secondary malignant tumors or other tumors within 3 years before the start of the study and there is metastasis of the brain or meninges.
10. Researchers believe that their compliance is poor
11. There are contraindications for Apatinib and S-1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-08-10 (Estimated); Study Completion 2020-08-10 (Estimated)

PRIMARY OUTCOMES:
PFS | 12 month after first treatment
  progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: xiao qing Jiang, professor, Principal Investigator — 700 Moyu Road North, Jiading District,Eastern Hepatobiliary Surgery Hospital, Shanghai, China
Locations (1):
- xiao qing xiao qing Jiang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No